CLINICAL TRIAL: NCT04210180
Title: Combination of E-cigarettes and Varenicline for Tobacco Harm Reduction
Acronym: EVAR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rose Research Center, LLC (Industry)
Collaborators: Foundation for a Smoke Free World INC (Other)
Responsible Party: Principal Investigator, Jed Rose, President and CEO, Rose Research Center, LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVAR
Record Dates: First submitted 2019-12-04; First posted 2019-12-24 (Actual); Results first posted 2022-02-08 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Smoking Cessation; Harm Reduction
MeSH Terms: conditions — Smoking Cessation; Harm Reduction | interventions — Varenicline; Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Varenicline plus e-cigarette (Experimental): Participants enrolled in the study will receive a G6 e-cigarette at V2 for ad libitum use. The FDA approved starter kit of varenicline will be provided to participants at V3 (0.5 mg nightly for days 1-3, then 0.5 mg twice daily for days 4-7) along with additional G6 cartomizers. After the first week of varenicline, participants will receive the FDA-approved standard dose of varenicline (1 mg twice daily) and will continue to receive enough G6 cartomizers for the next 11 weeks.
  Interventions: Drug: Varenicline; Other: e-cigarette

INTERVENTIONS:
Drug: Varenicline — 0.5 mg nightly for days 1-3, then 0.5 mg twice daily for days 4-7; then 1 mg twice daily for the remaining 11 weeks.
  Other Names: Chantix
Other: e-cigarette — Each G6 prefilled cartomizer contains a 50/50 blend nicotine salt with 35mg nicotine strength.
  Other Names: Halo G6

SUMMARY:
This open-label study will explore the impact of varenicline on the process of switching from combustible cigarettes (CC) to an e-cigarette. Varenicline is currently the most efficacious single pharmacotherapy for smoking cessation, and through its actions as an agonist or partial agonist at various nicotinic acetylcholine receptor subtypes, serves to diminish the rewarding effects of cigarette smoking. Diminishing the rewarding effects of smoking might facilitate the transition from CC to e-cigarettes. On the other hand, varenicline might attenuate the rewarding effects of nicotine-containing e-cigarettes as well, which could hamper the transition. Thus, the study will provide important information about the actions of varenicline on CC as well as e-cigarettes. There is no therapeutic intent in that smokers' nicotine/tobacco dependence will not be treated; the goal is to switch from one form of nicotine/tobacco dependence (CC) to dependence on a different tobacco product (e-cigarettes).

ELIGIBILITY:
Inclusion Criteria:

1. Has signed the ICF and is able to read and understand the information provided in the consent form.
2. Is 21 to 65 years of age (inclusive) at screening.
3. Smokes at least 10 commercially available cigarettes per day (no brand restrictions), for the last 12 months.
4. Has an expired air carbon monoxide reading of at least 10 ppm at screening.
5. Interested in switching to an electronic cigarette.
6. Willing and able to comply with the requirements of the study.
7. Owns a smart phone with text message and data capabilities compatible with necessary surveys.

Exclusion Criteria:

1. Is unhealthy or cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason) as judged by the Investigator or designated medical staff based on all available assessments from the screening period (e.g., safety laboratory, vital signs, physical examination, Ankle-Brachial Index, ECG, concomitant medications and medical history).
2. PHQ-9 score greater than 9, or a score greater than 0 on item #9 ("Thoughts that you would be better off dead, or of hurting yourself in some way") at screening.
3. Planned use of an FDA-approved smoking cessation product during the study.
4. High blood pressure (systolic > 150 mmHg or diastolic >95 mmHg) at screening.
5. Body mass index (BMI) less than 15.0 kg/m2 or greater than 40.0 kg/m2.
6. Coronary heart disease, structural cardiac disease (including, but not limited to valvular heart disease or cardiac murmurs), cardiac dysrhythmias, syncope, cardiac chest pain, or history of heart attack or heart failure.
7. Has received psychotherapy or behavioral treatments potentially impacting symptoms of depression, anxiety, or nicotine withdrawal within 30 days of screening, or during the study.
8. Taking antidepressants, psychoactive medications (e.g. antipsychotics, benzodiazepines, hypnotics) or medications that prolong QTc.
9. Use of any of these products in the past 30 days: a. Illegal drugs (or if the urine drug screen is positive for cocaine, THC, amphetamines, methamphetamines, or opiates); b. Experimental (investigational) drugs that are unknown to subject; c. Chronic opiate use.
10. Use of smokeless tobacco (chewing tobacco, snuff), cigars (except for "Black & Mild" cigars or Cigarillos), pipes, hookah, e-cigarettes, nicotine replacement therapy or other smoking cessation treatments within 14 days of screening.
11. Pregnant or nursing (by self-report) or has a positive pregnancy test.
12. Enrollment requirements met.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Rose Research Center, Charlotte, North Carolina
  - Rose Research Center, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in both the Raleigh, NC and Charlotte, NC offices of Rose Research Center. Enrollment started on 19 Nov 2019 and ended on 08 Jul 2020.
Period: Overall Study
Arm/Group | Varenicline Plus E-cigarette
Started | 25
Completed | 23
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline Plus E-cigarette
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.92 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participant Reporting Continuous Complete Switching From Cigarettes to Halo G6
Description: The primary switching outcome will be smoking abstinence during weeks 8-11 post-switching date. Complete switching from combustible cigarette use at each time point will be defined by a self-report of no cigarette smoking (not even a puff) since the prior session.
Time Frame: Weeks 8-11
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Plus E-cigarette
Number analyzed (Participants) | 25
Participants | 8

2. Primary Outcome: Number of Participants Confirmed (by Expired Air CO) to Have Switched From Cigarettes to Halo G6
Description: The primary switching outcome will be smoking abstinence during weeks 8-11 post-switching date. Complete switching from combustible cigarette use at each time point confirmed by an expired air CO reading of less than 5 ppm.
Time Frame: Weeks 8-11
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Plus E-cigarette
Number analyzed (Participants) | 25
Participants | 8

3. Secondary Outcome: Number of Participants Reporting Point Abstinence From Smoking Cigarettes at 6 Months Post-Switch
Description: Point abstinence will be defined by a self-report of no cigarette smoking (not even a puff) in the last seven days at six months post-switch.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Varenicline Plus E-cigarette
Number analyzed (Participants) | 25
Participants | 16

4. Other Pre Specified Outcome: Mean Changes in Arterial Flow When Smokers Switch From Cigarettes to E-cigarettes
Description: Ankle-Brachial Index (ABI) use to evaluate vascular changes when smokers change from cigarettes to e-cigarettes over a 13-week period. Measurements will be obtained using a manual sphygmomanometer and an 8- to 10- MHz doppler ultrasound probe. Subjects will undergo this testing at Visit 1 (baseline data) and at the end of study (Visit 7).
  Ankle Brachial Index (ABI) is the ratio of the blood pressure in the lower legs to the blood pressure in the arms. The normal range for the ankle-brachial index is between 0.90 and 1.30. An index of 0.41 to 0.90 indicates mild to moderate arterial disease and an index of 0.40 and lower indicates severe disease
Time Frame: Baseline (Visit 1) and 13 weeks (Visit 7)
Population: 10 participants were not able to come to the lab for ABI evaluation at Visit 7 because of COVID restrictions.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Varenicline Plus E-cigarette
Number analyzed (Participants) | 13
ratio | -0.05 (0.12)

ADVERSE EVENTS:
Time Frame: Data were collected during the 13 week study period.
Arm/Group | Varenicline Plus E-cigarette
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 1/25
Other Adverse Events (participants affected / at risk) | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Plus E-cigarette (N=25)
Allergic Reaction to lidocaine (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscular weakness caused by interarticular joint injection, requiring hospitalization, self-resolved within 48 hours.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline Plus E-cigarette (N=25)
Vomiting (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 6 (6)
Insomnia (Nervous system disorders) | 4 (5)
Nightmares/ Vivid Dreams (Nervous system disorders) | 3 (3)
Agitation/Anxiety (Psychiatric disorders) | 2 (2)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT04210180/Prot_SAP_000.pdf